CLINICAL TRIAL: NCT06376214
Title: Daratumumab and Dexamethasone Combined With Pomalidomide (DPD) or ASCT in the Treatment of Newly Diagnosed Systemic Light Chain Amyloidosis (AL Amyloidosis): a Prospective, Single Center Clinical Trial
Brief Title: Daratumumab for Patients With Light Chain Amyloidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhi-Hong Liu, MD, Professor, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02
Record Dates: First submitted 2024-03-29; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Light Chain (AL) Amyloidosis
Keywords: light chain amyloidosis; daratumumab; stem cell transplantation
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — Hyaluronoglucosaminidase; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- long-term daratumumab treatment group (group A) (Active Comparator): The patient will receive the standard protocol of daratumumab combined with dexamethasone treatment, once a week for the first two months, once every two weeks for four months, and then once a month for 18 months.
  Interventions: Drug: Dratumumab / Hyaluronidase Injection [Darzalex Faspro]
- daratumumab combine with ASCT treatment group (group B) (Experimental): This group of patients will first receive two courses of treatment with the standard protocol of daratumumab combined with dexamethasone. Subsequent patients will receive ASCT treatment, and patients who achieve VGPR or CR after transplantation treatment will be followed up for observation
  Interventions: Drug: Dratumumab / Hyaluronidase Injection [Darzalex Faspro]; Procedure: autologous stem cell transplantation (ASCT)
- Daratumumab and Dexamethasone combined with pomalidomide (DPD) (group C) (Experimental): newly diagnosed stage IIIb AL amyloidosis patients will received Daratumumab (16mg/kg), dexamethasone (40mg) and pomalidomide. The usage of Daratumumab and dexamethasone is the same as group A. Patients received oral pomalidomide on days 1-21 of a 28-days cycle from cycle 1 to 6. The dose of pomalidomide is adjusted based on the patient's renal function and ECOG score.
  Interventions: Drug: Dratumumab / Hyaluronidase Injection [Darzalex Faspro]; Drug: Pomalidomide 4 MG

INTERVENTIONS:
Drug: Dratumumab / Hyaluronidase Injection [Darzalex Faspro] — Daratumumab will be administered at the FDA-approved dose of 16mg/kg as an intravenous infusion.
  Other Names: DARA
Drug: Pomalidomide 4 MG — Patients received oral pomalidomide on days 1-21 of a 28-days cycle from cycle 1 to 6.
  Arms: Daratumumab and Dexamethasone combined with pomalidomide (DPD) (group C)
Procedure: autologous stem cell transplantation (ASCT) — The ASCT protocol included mobilisation with colony-stimulating factor alone and conditioning with high-dose melphalan140-200 mg/m2
  .
  Arms: daratumumab combine with ASCT treatment group (group B)

SUMMARY:
This is a prospective, single-center study exploratory clinical trial, aim to exploring the efficacy and safety of daratumumab in patients with AL amyloidosis, patients were divided into three groups: one group received long-term treatment with daratumumab based regimen, and the other group received autologous stem cell transplantation after two standard treatment courses with daratumumab based regimen, and the third group consists of newly diagnosed stage IIIb AL amyloidosis patients who plan to receive DPD treatment. The purpose of this study is to observe the efficacy and safety of Daratumumab, in the treatment of newly diagnosed systemic AL amyloidosis.

DETAILED DESCRIPTION:
This is a prospective, single-center study exploratory clinical trial, aim to exploring the efficacy and safety of daratumumab in patients with AL amyloidosis, patients were divided into three groups: one group received long-term treatment with daratumumab based regimen (group A) and the other group received autologous stem cell transplantation after two standard treatment courses with daratumumab based regimen (group B) , and the third group consists of newly diagnosed stage IIIb AL amyloidosis patients who plan to receive DPD treatment (group C). Participants with AL Amyloidosis will receive the drug daratumumab by IV infusion once weekly for two months, then every 2 weeks for four months, then once each month. Study treatment may continue until disease progression, unacceptable toxicity, or decision to withdraw from the trial. Disease evaluations will be performed every three months until disease progression. Group C were given Daratumumab (16mg/kg), dexamethasone (40mg) and pomalidomide. The usage of Daratumumab and dexamethasone is the same as group A and B. Patients received oral pomalidomide on days 1-21 of a 28-days cycle from cycle 1 to 6. The dose of pomalidomide is adjusted based on the patient's renal function and ECOG score.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged ≥18 and ≤75 years;
2. Newly diagnosed AL amyloidosis ((confirmed by pathological examination with at least one major organ involvement (heart, kidney, or liver));
3. In group A and B, according to the Mayo 2004 staging system, the disease is classified as stage Ⅰ-ⅢA; In group C, according to the Mayo 2004 staging system, the disease is classified as stage IIIB: NT⁃proBNP>8500ng/L and cTnT>0.035μg/L or cTnI>0.01g/L;
4. Participants must personally sign an informed consent form approved by the Ethics Committee before the start of the study;
5. Expected survival ≥ 12 weeks;
6. ECOG performance status≤ 2;
7. Female participants of childbearing potential must agree to use effective contraception from the day of signing the informed consent until 365 days after the infusion. Effective contraception is defined as abstinence or the use of a contraceptive method with a failure rate of <1% per year.

Exclusion Criteria:

1. eGFR< 30ml/min/1.73m2;
2. Combined multiple myeloma;
3. Acute or chronic infection requiring treatment within 30 days prior to baseline;
4. Pregnant or breastfeeding women.
5. Participants known to have life-threatening allergic reactions, hypersensitivity, or intolerance to Monoclonal antibodies or immune modulators.
6. Other conditions deemed by the researcher as unsuitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hematological complete response rate | 6 months
  the 6 months overall hematologic complete response rate after treatment.
Organ response rate | 1 year
  the 1-year organ response rate after treatment

SECONDARY OUTCOMES:
Time to Next Treatment | 3 years
  Number of months from study drug initiation to starting another treatment
Progression-free survival | 3 years
  the 3 years progression-free survival after treatment
Overall survival | 5 years
  the 5 years overall survival after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xianghua Huang, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- National Clinical Research Center for Kidney Diseases, Jinling Hospital, Nanjing, Jiangsu, China